CLINICAL TRIAL: NCT06409273
Title: Effect of Hybrid Versus Face-to-face Teaching on Course Assessment and Evaluation in Postgraduate General Practice Students: a Randomized Controlled Trial
Brief Title: Hybrid Course Assessment and Evaluation
Acronym: HOME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HOME
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Education, Medical
Keywords: Medical education; Students; dissertations, academic; Evaluation studies; Educational measurement

STUDY DESIGN:
Intervention Model Description: Mixed-methods study
  1. Single-blind, randomized, controlled trial with two 1:1 parallel arms
  2. Qualitative analysis of open-ended questions in a questionnaire
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Hybrid course : asynchronous online interactive course (2h30, 45%) followed by face-to-face socio constructivist teaching (3h00, 55%)
  Interventions: Other: Hybrid course on medical thesis for post graduates general practice students
- Control (Active Comparator): Face-to-face socio constructivist teaching (100%) (5h30)
  Interventions: Other: Face-to-face teaching on medical thesis for post graduates general practice students

INTERVENTIONS:
Other: Hybrid course on medical thesis for post graduates general practice students — Students randomised to the intervention group will log on to interactive online teaching for a maximum time of 2.5 hours, and then follow face-to-face socio-constructivist teaching in small groups (n=22 max), building on the knowledge they have acquired. The aim of this peer-to-peer face-to-face teaching is to develop problem-solving skills.
  Arms: Intervention
Other: Face-to-face teaching on medical thesis for post graduates general practice students — Students randomised to the control group will be taught entirely face-to-face in small groups (n=22 max). The course duration and teaching objectives are identical to those of the intervention group. Student consent and randomization will be carried out on the morning of the course to avoid contamination and attrition bias.
  Arms: Control

SUMMARY:
The academic training of French postgraduate students in general practice (E3CMG) is facing a challenge due to the increasing gap between the number of students and the available teaching hours. To accommodate the growing number of students, asynchronous acquisition of knowledge prior to a reduced face-to-face teaching would maintain the capacity to provide socio-constructivist teaching useful for developing problem-solving skills (i.e. thesis design and feasibility assessment). The main objective of this randomized controlled trial is to evaluate the effect of hybrid versus face-to-face socio-constructivist teaching on French E3CMG course assessment and evaluation.

DETAILED DESCRIPTION:
The E3CMG will be invited to attend one of the two teaching days in accordance with the usual university procedure. They will be gathered in an amphitheater at the start of the teaching session (9:00 a.m.), where they will receive oral and written information about the study. Blocked randomization with randomly selected block sizes will be performed among students who have signed a written consent to participate in the study. Non-participants in the study will be assigned to one of the two teaching formats without randomization and respecting the need to achieve close class sizes. Their teaching assessments will not be extracted and analyzed as part of the study.

This late randomization procedure makes it possible to

* allow students to change teaching day without regard to the study
* avoid contamination bias caused by some students accessing the asynchronous interactive course before class
* ensure compliance with the study protocol (systematic access to the asynchronous interactive course by students in the intervention group)
* Control the time spent on the asynchronous interactive course to ensure that the time spent by students actually corresponds to that stated in the protocol.
* To limit missing data management procedures: data collection on the day of teaching, and randomization only of students present on the day of teaching (limits attrition bias).

The 4 teachers on the first teaching day will be randomly assigned to the groups (May 14). If they take part in the second teaching day (05/21), they will teach in the other group in order to minimize a bias in the evaluation of the main judgment criterion linked to teacher quality.

The study begins on May 14, 2024 or May 21, 2024, depending on the participant's assigned teaching day, and ends on 11/14/2024. The maximum duration of participation in the study is therefore 6 months. The student's actual participation is 1 day, as data collection on 14/11 is automated and does not require any intervention by the participant.

No health data will be collected. Data will be collected via a self-administered questionnaire with a randomized order of questions at the end of the teaching day, and at 6 months via the university's database of thesis forms.

The number of participants to be included in the study is 72 per arm. This is necessary to demonstrate a difference in the primary endpoint of 10%, with a standard deviation of 4 points, an alpha risk of 5%, and a statistical power of 85%, for a two-tailed t-test of comparison of observed means. The theoretical maximum number of students included in the study was 83 per group, allowing for a 13% refusal rate (n=22 students).

A two-sided superiority test will be conducted, with a multivariate analysis and sensitivity analysis. To account for multiple comparisons regarding secondary objectives, a fixed sequence procedure will be performed. Once one hypothesis is tested and found to be not significantly different from the null hypothesis, all subsequent tests and results will be considered as explanatory. The secondary objectives described below are classified according to this procedure.

ELIGIBILITY:
Inclusion Criteria:

• Postgraduate general practice students registered for assessed course.

Exclusion Criteria:

• Unsigned written consent to participate after oral and written information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-05-14 (Estimated); Primary Completion 2024-05-21 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
Self-assessment score for learning outcomes | At the end of the teaching day
  Sum of self-assessment score for knowledge (10 points) and self-assessment score for skills (10 points). Maximum value = 20, Minimum Value = 0. Higher score means a better outcome.

SECONDARY OUTCOMES:
Overall satisfaction score | At the end of the teaching day
  Sum of the satisfaction score for knowledge-related learning objectives (satisfaction score 1, 10 points) and the satisfaction score for skill-related learning objectives (satisfaction score 2, 10 points). Maximum value = 20, Minimum Value = 0. Higher score means a better outcome.
Self-assessment score for knowledge (10 points) | At the end of the teaching day
  10-point score based on a questionnaire completed by students to assess knowledge acquisition. Maximum value = 10, Minimum Value = 0. Higher score means a better outcome.
Self-assessment score for skills (competencies) (10 points) | At the end of the teaching day
  10-point score based on a questionnaire completed by students to assess problem-solving skills acquisition. Maximum value = 10, Minimum Value = 0. Higher score means a better outcome.
Satisfaction score 1 | At the end of the teaching day
  10-point score for student satisfaction regarding knowledge-related learning objectives. Maximum value = 10, Minimum Value = 0. Higher score means a better outcome.
Satisfaction score 2 | At the end of the teaching day
  10-point score for student satisfaction regarding skills-related learning objectives. Maximum value = 10, Minimum Value = 0. Higher score means a better outcome.
Submitting a thesis form | 6 months after the course
  A thesis form is a document submitted by students to the university department of general medicine for proofreading before validation concerning the problematization and feasibility of the project. The course evaluated is likely to improve the time taken to submit the thesis form.

CONTACTS AND LOCATIONS:
Overall Officials: Rémy Boussageon, MD, PhD, Study Chair — Lyon 1 University & LBBE UMR 5558, CNRS; Marion Lamort-Bouché, MD, PhD, Study Director — Research on Healthcare Performance Lab U1290, Inserm; Pierre-Yves Meunier, MD, Principal Investigator — University Lyon 1; Sophie Schlatter, PhD, Study Chair — Research on Healthcare Performance Lab U1290, Inserm

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest on medical education. Data or samples shared will be coded.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted immediatly after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Approval of the request by Pierre-Yves Meunier (principal investigator) and Marion-Lamort Bouché (study director) and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party. For more information or to submit a request, please contact pierre-yves.meunier@univ-lyon1.fr